CLINICAL TRIAL: NCT06918392
Title: Field-test and Psychometric Validation of the Pectus Excavatum Evaluation Questionnaire in the Dutch Pectus Excavatum Population
Acronym: TRANSLATE
Status: Not yet recruiting | Type: Observational
Sponsor: Zuyderland Medisch Centrum (Other)
Responsible Party: Principal Investigator, Erik de Loos, Principal Investigator, Zuyderland Medisch Centrum
Other Study IDs: METCZ20210182
Record Dates: First submitted 2025-03-24; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Pectus Excavatum
MeSH Terms: conditions — Funnel Chest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pectus excavatum patients: pectus excavatum patients aged 12 to 18 years old who are scheduled for a Nuss procedure, and their parents or legal guardians.

SUMMARY:
A questionnaire that can measure disease severity from the patients perspective in patients with pectus excavatum already exists in English (Pectus Excavatum Evaluation Questionnaire; PEEQ). This questionnaire was recently translated into Dutch. Before this Dutch version can be used, it needs to be tested by a number of patients.

Data will be collected at three moments:

1. Preoperatively: The PEEQ will be completed on paper during the outpatient clinic visit.
2. Postoperatively: The PEEQ will be completed electronically 2 months post-surgery.
3. Test-retest reliability: The PEEQ will be administered electronically at least two weeks after a previous assessment.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants will be pectus excavatum patients aged 12 to 18 years old who are scheduled for a Nuss procedure. Parents or legal guardians will also be invited to complete the parent section of the PEEQ.

Exclusion Criteria:

* Exclusion criteria will be the inability of the patient or their parent/guardian to complete the corresponding section of the questionnaire due to language barriers.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants will be identified and enrolled during their preoperative visit at the outpatient clinic of Zuyderland Medical Center by a member of the research team.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Structural validity | Pre-operative assessment of pectus excavatum evaluation questionnaire at the outpatient clinic visit. Minimum score of this questionnaire is 22, maximum score is 88, a higher score indicates a lower disease-related quality of life.
  A Kaiser-Meyer-Olkin (KMO) test and Bartlett's test of sphericity are performed to assess the adequacy of patient sampling before performing further structural tests. Threshold values of ≥ 0.70 in KMO test and p < 0.05 in Bartlett's test of sphericity indicate the suitability of the collected data for factor analysis (6,7). Exploratory factor analysis (EFA), using principal axis factoring and a promax rotation method, will be conducted to identify the underlying factor structure for both the child and parent sections (8,9). These factor structures will later be subjected to confirmatory factor analysis (CFA), using polychoric correlations and robust maximum likelihood estimation, to evaluate the validity of the structures derived from EFA (8,10). Within EFA, the Kaiser criterion (eigenvalue > 1), explained variance (≥50%), and interpretability principle will be applied to determine the number of factors to be retained. Squared multiple correlations are used to compute the communality
Internal consistency | Pre-operative assessment of pectus excavatum evaluation questionnaire at the outpatient clinic visit. Minimum score of this questionnaire is 22, maximum score is 88, a higher score indicates a lower disease-related quality of life.
  Cronbach's alpha coefficient, a measure of internal consistency, will be calculated for each subscale. A value > .70 indicates sufficient reliability of the questionnaire for application at the group level, while a value > .90 implies suitability for individual assessment
Test-retest reliability | Pre-operative assessment of pectus excavatum evaluation questionnaire OR the 2 months postoperative assessment will be used as a baseline. Another assessment wil be performed minimally 2 weeks after one of the aforementioned assessments.
  Test-retest reliability for each subscale will be evaluated using a two-way mixed-effects model for the intraclass correlation coefficient (ICC), type (3.1), with 95% confidence intervals reported (CI) (15). The strength of agreement will be interpreted following the guideline provided by Cicchetti (1994) (16): < 0.40 = poor, 0.40-0.59 = fair, 0.60-0.74 = good, 0.75-1.00 = excellent. For individual items, quadratic weighted Cohen's kappa will be calculated along with its 95% to identify problematic items, with interpretation based on the standards proposed by Landis and Koch (1977) (17): <0 = poor, 0.01-0.20 = slight, 0.21-0.40 = fair, 0.41-0.60 = moderate, 0.61-0.80 = substantial, and 0.81-.001 = almost perfect.
Responsiveness | re-operative assessment of pectus excavatum evaluation questionnaire at the outpatient clinic visit. Minimum score of this questionnaire is 22, maximum score is 88, a higher score indicates a lower disease-related quality of life.
  The responsiveness of the questionnaire will be determined using the construct approach in which preoperative and postoperative scores are compared using a paired t-test or Wilcoxon signed-rank test for skewed data. The effect size will be expressed in Cohen's d and is calculated as the mean difference divided by the standard deviation of the difference. We hypothesize that the total score on the PEEQ and mean scores per subscale improve after surgical correction of the pectus excavatum deformity as demonstrated by the original questionnaire (2,3). Responsiveness of individual items will be evaluated using a paired t-test or Wilcoxon signed-rank test, as appropriate, to guide further item refinement.
Smallest detectable change | Pre-operative assessment of pectus excavatum evaluation questionnaire and two months postoperative assessment. Minimum score of this questionnaire is 22, maximum score is 88, a higher score indicates a lower disease-related quality of life.
  The standard error of measurement (SEM) quantifies the precision of the scores across different time points and is calculated as (18):
  SEM = squareroot of MSE
  Where:
  · Mean square error (MSE) is the error term obtained from repeated measures ANOVA
  The SDC represents the minimum change in points a patient must score on the questionnaire over time to ensure the observed change reflects a real change and not a measurement error. The SDC is expressed in points on the PEEQ and will be calculated for the mean scores per subscale, and the total scores of the child's section, parent's section and entire questionnaire. The SDC at a 95% confidence level will be calculated as (18):
  SDC = 1.96 x square root of 2 x SEM
  Where:
  * 1.96 is the z-score corresponding to a 95% confidence level
  * square root of 2 x SEM accounts for the error variance from both time points

SECONDARY OUTCOMES:
Floor and ceiling effects | Pre-operative assessment of pectus excavatum evaluation questionnaire and two months postoperative assessment. Minimum score of this questionnaire is 22, maximum score is 88, a higher score indicates a lower disease-related quality of life.
  The floor and ceiling effects will be assessed by calculating the proportion of participants scoring the lowest or highest possible scores. Effects are considered substantial if > 15% of the participants score at the extremes for a specific item or subscale (18).

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: trough publication in a peer-reviewed journal

REFERENCES:
- [Background] Janssen N, Daemen JHT, van Polen EJ, Coorens NA, Jansen YJL, Franssen AJPM, Hulsewe KWE, Vissers YLJ, Haecker FM, Milanez de Campos JR, de Loos ER; Chest Wall International Group Collaborator Group. Pectus Excavatum: Consensus and Controversies in Clinical Practice. Ann Thorac Surg. 2023 Jul;116(1):191-199. doi: 10.1016/j.athoracsur.2023.02.059. Epub 2023 Mar 29. PMID 36997016
- [Background] Terwee CB, Bot SD, de Boer MR, van der Windt DA, Knol DL, Dekker J, Bouter LM, de Vet HC. Quality criteria were proposed for measurement properties of health status questionnaires. J Clin Epidemiol. 2007 Jan;60(1):34-42. doi: 10.1016/j.jclinepi.2006.03.012. Epub 2006 Aug 24. PMID 17161752
- [Background] Landis JR, Koch GG. The measurement of observer agreement for categorical data. Biometrics. 1977 Mar;33(1):159-74. PMID 843571
- [Background] Cicchetti D V. Guidelines, criteria, and rules of thumb for evaluating normed and standardized assessment instruments in psychology. Psychol Assess. 1994;6:284-90.
- [Background] Shrout PE, Fleiss JL. Intraclass correlations: uses in assessing rater reliability. Psychol Bull. 1979 Mar;86(2):420-8. doi: 10.1037//0033-2909.86.2.420. PMID 18839484
- [Background] Fayers PM. Quality of life : The assessment, analysis, and reporting of patient-reported outcomes. 3rd ed. Chichester: Wiley Blackwell; 2016.
- [Background] Schreiber JB, Nora A, Stage FK, Barlow EA, King J. Reporting Structural Equation Modeling and Confirmatory Factor Analysis Results: A Review. J Educ Res. 2006;99:323-38
- [Background] Kline P. An Easy Guide to Factor Analysis. 1st ed. New York: Routledge; 2014.
- [Background] Pituch KASJ. Applied multivariate statistics for the social sciences: Analyses with SAS and IBM's SPSS. 6th ed. New York: Routledge; 2016.
- [Background] Holgado-Tello FP, Chacón-Moscoso S, Barbero-García I, Vila-Abad E. Polychoric versus Pearson correlations in exploratory and confirmatory factor analysis of ordinal variables. Qual Quant. 2010;44:153-66.
- [Background] Osborne JW, Costello AB. Best practices in exploratory factor analysis: four recommendations for getting the most from your analysis. Practical assessment, research and evaluation. 2005;10:1-9.
- [Background] Brown T. Confirmatory factor analysis for applied research. 2nd ed. New York: Guilford Press; 2015.
- [Background] Hoelzle JB, J. Meyer G. Exploratory Factor Analysis: Basics and Beyond. In: Handbook of Psychology, 2nd ed. New York: Wiley; 2012.
- [Background] Watkins MW. Exploratory Factor Analysis: A Guide to Best Practice. Journal of Black Psychology. 2018;44:219-46.
- [Background] Mokkink L, Prinsen C, Patrick D, et al. COSMIN Study Design checklist for Patient-reported outcome measurement instruments. 2019. Available online: https://www.cosmin.nl/wp-content/uploads/COSMIN-study-designing-checklist_final.pdf.
- [Background] Janssen N, Daemen JHT, van Polen EJ, Jansen YJL, Hulsewe KWE, Vissers YLJ, de Loos ER. Translation, cultural adaptation and linguistic validation of the pectus excavatum evaluation questionnaire. J Thorac Dis. 2022 Jul;14(7):2556-2564. doi: 10.21037/jtd-22-252. PMID 35928622
- [Background] Kelly RE Jr, Cash TF, Shamberger RC, Mitchell KK, Mellins RB, Lawson ML, Oldham K, Azizkhan RG, Hebra AV, Nuss D, Goretsky MJ, Sharp RJ, Holcomb GW 3rd, Shim WK, Megison SM, Moss RL, Fecteau AH, Colombani PM, Bagley T, Quinn A, Moskowitz AB. Surgical repair of pectus excavatum markedly improves body image and perceived ability for physical activity: multicenter study. Pediatrics. 2008 Dec;122(6):1218-22. doi: 10.1542/peds.2007-2723. PMID 19047237
- [Background] Lawson ML, Cash TF, Akers R, Vasser E, Burke B, Tabangin M, Welch C, Croitoru DP, Goretsky MJ, Nuss D, Kelly RE Jr. A pilot study of the impact of surgical repair on disease-specific quality of life among patients with pectus excavatum. J Pediatr Surg. 2003 Jun;38(6):916-8. doi: 10.1016/s0022-3468(03)00123-4. PMID 12778393
- [Background] Mohamed JS, Tan JW, Tam JKC. Quality of life with minimally invasive repair of pectus excavatum: a systematic review and meta-analysis. Ann Transl Med. 2023 Dec 20;11(12):407. doi: 10.21037/atm-23-1647. Epub 2023 Dec 6. PMID 38213813
- [Derived] Janssen N, van Polen EJ, Daemen JHT, Franssen AJPM, Winkens B, Hulsewe KWE, Vissers YLJ, de Loos ER. Protocol for the field-test and psychometric validation of the pectus excavatum evaluation questionnaire in the Dutch pectus excavatum population. Transl Pediatr. 2025 Apr 30;14(4):694-699. doi: 10.21037/tp-2024-616. Epub 2025 Apr 27. PMID 40386365